CLINICAL TRIAL: NCT05614544
Title: A 2-Part, Dose-Finding and Human Abuse Potential Study Of HSK3486 Injection In Nondependent, Recreational Central Nervous System Depressant Users
Brief Title: Dose-Finding and Human Abuse Potential Study Of HSK3486 Injection In Nondependent, Recreational Central Nervous System Depressant Users
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Haisco-USA Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSK3486-110
Record Dates: First submitted 2022-10-12; First posted 2022-11-14 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2022-10

CONDITIONS: General Anesthesia
MeSH Terms: interventions — HSK3486; Propofol

STUDY DESIGN:
Who Masked: Participant
Masking Description: double-blind, placebo- and active-controlled 4 period, 4 way crossover design to assess the abuse potential of HSK3486
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Treatment A: HSK3486 dose 1 (Experimental): Treatment A: HSK3486 dose 1 (IV bolus over 30 seconds [+5 seconds] from a syringe; dose to be determined in Part 1)
  Interventions: Drug: HSK3486
- Treatment B: HSK3486 dose 2 (Experimental): Treatment B: HSK3486 dose 2 (IV bolus over 30 seconds [+5 seconds] from a syringe; dose to be determined in Part 1)
  Interventions: Drug: HSK3486
- Treatment C: Propofol (Active Comparator): Treatment C: Propofol (IV bolus over 30 seconds [+5 seconds] from a syringe; dose to be determined in Part 1)
  Interventions: Drug: Propofol
- Treatment D: Placebo (Placebo Comparator): Treatment D: Placebo (Treatment A matched) (IV bolus over 30 seconds [+5 seconds] from a syringe)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HSK3486 — HSK3486 for induction of general anesthesia
  Arms: Treatment A: HSK3486 dose 1; Treatment B: HSK3486 dose 2
Drug: Propofol — Propofol for induction of general anesthesia
  Arms: Treatment C: Propofol
Drug: Placebo — Intralipid
  Arms: Treatment D: Placebo

SUMMARY:
Part 1: To determine the doses of IV HSK3486 and propofol for use in Part 2, the abuse potential part of the study.

Part 2: To evaluate the abuse potential of HSK3486 compared with propofol when administered IV to healthy nondependent, recreational CNS depressant drug users.

DETAILED DESCRIPTION:
This single center study will consist of 2 parts. Part 1 will be an open-label, dose-finding study of HSK3486 and propofol conducted in up to 48 recreational users of CNS depressants to determine the appropriate doses to be used in Part 2 of the study. Part 2 will be a randomized, double-blind, placebo- and active-controlled 4-period, 4 way crossover, in approximately 42 healthy volunteers with prior recreational CNS depressant exposure. Both Part 1 and Part 2 of the study will consist of an outpatient Screening Visit, an in-clinic Treatment Phase, and Follow-up; Part 2 will also include a Qualification Phase.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to participate in the study, give written informed consent, and comply with the study restrictions.
2. Gender: male or female; females may be of childbearing potential, of nonchildbearing potential, or postmenopausal.
3. Age: 18 years to 55 years, inclusive, at Screening.
4. Body mass index (BMI): 18.0 kg/m2 to 30.0 kg/m2, inclusive.
5. Weight: ≥50 kg, inclusive.
6. Healthy subject, defined by the absence of evidence of any clinically significant, in the opinion of the Investigator, active or chronic disease following a detailed medical and surgical history, a complete physical examination including vital signs, 12-lead ECG, hematology, blood chemistry, serology, and urinalysis.
7. Subject must be a nondependent, nontreatment-seeking recreational CNS depressant user, defined as follows:

   * ≥10 lifetime nontherapeutic experiences (i.e., for psychoactive effects) with CNS depressants (e.g., benzodiazepines, barbiturates, opiates, zolpidem, zopiclone, propofol/fospropofol, gamma-hydroxybutyrate).
   * ≥1 nontherapeutic use of a CNS depressant within the 8 weeks prior to Screening.
   * ≥1 nontherapeutic use of benzodiazepines within the 12 months prior to Screening.
8. Ability and willingness to abstain from alcohol-, caffeine-, and xanthine-containing beverages or food (e.g., coffee, tea, cola, chocolate, energy drinks) from 48 hours (2 days) prior to first admission to the CRU, throughout the entire study, and until discharge.
9. All values for hematology and clinical chemistry tests of blood and urine within the normal range or show no clinically relevant deviations, as judged by the Investigator.
10. Females of childbearing potential, and males with female partner(s) of childbearing potential, as judged by the Investigator, must agree to use 2 forms of contraception, 1 of which must be a barrier method, during the study and for 90 days after the last drug administration. Acceptable barrier forms of contraception are condom, cervical cap, and diaphragm. Acceptable non barrier forms of contraception for this study are an intrauterine device (IUD) including hormonal IUDs, oral contraceptives (used for ≥30 days prior to dosing any study treatment), and/or spermicide.
11. For females: a negative pregnancy test at Screening and Admission.
12. Postmenopausal females: defined as 12 months with no menses prior to Screening and a serum follicle stimulating hormone (FSH) >40 IU/L at Screening.
13. All nonregular medication (including over-the-counter medication, health supplements, and herbal remedies such as St. John's Wort extract) must have been stopped at least 14 days prior to (the first) admission to the CRU. An exception is made for acetaminophen, which is allowed up to admission to the CRU.
14. All prescribed medication must have been stopped at least 30 days prior to (first) admission to the clinical research center. An exception is made for hormonal contraceptives, which may be used throughout the study.
15. Able to speak, read, and understand English sufficiently to allow completion of all study assessments.

Exclusion Criteria:

1. An employee of the Sponsor or research site personnel directly affiliated with this study or their immediate family member (defined as a spouse, parent, child, or sibling, whether biological or legally adopted).
2. Drug or alcohol dependence within the 2 years prior to Screening (except nicotine and caffeine), as defined by the Diagnostic and Statistical Manual of Mental Disorders, fourth edition, text revision (DSM IV TR), and/or has ever participated or plans to participate in a substance or alcohol rehabilitation program to treat their substance or alcohol dependence.
3. Opioid dependence as judged by the Investigator after a naloxone challenge.
4. Women who are pregnant, lactating, or planning to attempt to become pregnant during this study or within 90 days of last study drug administration.
5. Males with female partners who are pregnant, lactating, or planning to attempt to become pregnant during this study or within 90 days of last study drug administration.
6. Positive drug and alcohol screen (tetrahydrocannabinol [THC], morphine/opiates, methadone, oxycodone, phencyclidine, cocaine, amphetamines, methamphetamines, ecstasy, barbiturates, benzodiazepines, tricyclic antidepressants, and alcohol) at each admission to the CRU. For THC, subjects should ideally test negative. However, eligibility decision with regards to THC use will be considered on a case by case basis, at the discretion of the Investigator.
7. Treatment with an investigational drug or device within 5 times the elimination half-life, if known (e.g., a marketed product) or within 30 days (if the elimination half-life is unknown) prior to first drug administration or is concurrently enrolled in any research judged not to be scientifically or medically compatible with this study. An exception may be made for subjects who participated in Part 1 of the study.
8. History or presence of clinically significant abnormality (e.g., obstructive sleep apnea) as assessed by physical examination, medical history, ECG, vital signs, or laboratory values, which, in the opinion of the Investigator, would jeopardize the safety of the subject or the validity of the study results.
9. Any disease which, in the opinion of the Investigator, poses an unacceptable risk to the subjects.
10. Mallampati intubation score >2.
11. History of clinically significant drug allergy diagnosed by a physician. Confirmatory circumstances would include treatment with epinephrine or in an emergency department.
12. Any personal or family history of issues with succinylcholine, such as malignant hyperthermia or pseudocholinesterase deficiency.
13. History of allergy, adverse reaction (including significant agitation, etc.), or hypersensitivity to propofol, lidocaine, other injected anesthetic agents, or related drugs.
14. History of allergy to eggs, egg products, soybeans or soy products.
15. Heavy smoker (>20 cigarettes per day) and/or is unable to abstain from smoking and/or the use of prohibited nicotine-containing products (including e-cigarettes, pipes, cigars, chewing tobacco, nicotine topical patches, nicotine gum, or nicotine lozenges) from 2 hours prior to dosing until at least 4 hours postdose during the in clinic periods.
16. Routine or chronic use of more than 3000 mg of acetaminophen daily.
17. Strenuous activity (such as exercise), sunbathing, and contact sports within 48 hours (2 days) prior to admission to the CRU, during the study, and until after discharge in the last study period.
18. History of donation of more than 450 mL of blood within 60 days prior to dosing in the CRU or planned donation before 30 days has elapsed since last intake of study drug.
19. Plasma or platelet donation within 7 days of dosing and throughout the entire study.
20. Average intake of more than 14 units of alcohol per week (1 unit of alcohol equals approximately 250 mL of beer, 100 mL of wine, or 35 mL of spirits). Alcohol consumption will be prohibited 48 hours prior to first admission to the CRU and throughout the entire study until the Follow-up visit (including washout period).
21. Positive screening test for hepatitis B surface antigen (HBsAg), anti-hepatitis C virus (HCV) antibodies, or anti-HIV 1 and 2 antibodies.
22. History of peripheral vasculopathy, including Raynaud's phenomenon.
23. History of seizures, seizure disorder, or known electroencephalogram (EEG) abnormalities.
24. History of mental illness, which, in the opinion of the Investigator, would jeopardize the safety of the subject or the validity of the study results.
25. Subject with a history of clinically significant head injury, ongoing seizure disorder, chronic tics, or diagnosis or family history of Tourette's syndrome.
26. Subjects with a history of serious structural cardiac abnormalities, cardiomyopathy, serious heart rhythm abnormalities, coronary artery disease, advanced arteriosclerosis, symptomatic cardiovascular disease, hypertension, or other cardiac problems.
27. Any history of clinically significant suicidality as assessed by the Investigator based upon clinical history, source documents, or scores on the Columbia Suicide Severity Rating Scale (C-SSRS).
28. History or presence of clinically significant hepatic or renal disease.
29. History of hyperthyroidism.
30. Difficulty with venous access or unsuitable or unwilling to undergo catheter insertion.
31. Use of a cytochrome P450 (CYP)2D6-inhibiting drug or a serotonergic drug within 14 days prior to first drug administration in the Qualification Phase.
32. Consumption of any nutrients known to modulate CYP enzymes activity (e.g., grapefruit or grapefruit juice, pomelo juice, star fruit, or Seville [blood] orange products) within 14 days prior to administration of study medication and during the study (including washout period) until after discharge in the last study period.
33. A subject who, in the opinion of the Investigator or designee, is considered unsuitable or unlikely to comply with the study protocol for any reason.
34. A subject who has pending legal charges or is on probation.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2022-08-16 (Actual); Primary Completion 2023-10-03 (Actual); Study Completion 2023-10-03 (Actual)

PRIMARY OUTCOMES:
Part 1 | Screening between Day -28 and Day -5; confinement period 9 days in clinic from Day -4 (admission) to 24 hours after study drug administration in period 4; follow-up 3 to 7 days after study drug administration
  To determine the doses of IV HSK3486 and propofol for use in Part 2, the abuse potential part of the study
Part 2 | Screening between Day -28 and Day -2; confinement period 2 days in clinic from Day -1 (admission) to 24 hours after study drug administration; follow-up 3 to 7 days after study drug administration
  To evaluate the abuse potential of HSK3486 compared with propofol when administered IV to healthy nondependent, recreational CNS depressant drug users

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of HSK3486 in healthy, nondependent, recreational CNS depressant drug users | Screening between Day -28 and Day -5; confinement period 9 days in clinic from Day -4 (admission) to 24 hours after study drug administration in period 4; follow-up 3 to 7 days after study drug administration
  To evaluate the safety and tolerability of HSK3486 in healthy, nondependent, recreational CNS depressant drug users
• To evaluate the safety and tolerability of HSK3486 compared to propofol when administered IV to healthy nondependent, recreational CNS depressant drug users | Screening between Day -28 and Day -2; confinement period 2 days in clinic from Day -1 (admission) to 24 hours after study drug administration; follow-up 3 to 7 days after study drug administration
  * To evaluate the safety and tolerability of HSK3486 compared to propofol when administered IV to healthy nondependent, recreational CNS depressant drug users
  * To evaluate the PK profile of HSK3486 when administered IV to healthy nondependent, recreational CNS depressant drug users

CONTACTS AND LOCATIONS:
Locations (1):
- ICON (LPRA) - Salt Lake, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Undecided